CLINICAL TRIAL: NCT00053872
Title: A Prospective Randomised Controlled Trial Of Hyperfractionated Versus Conventionally Fractionated Radiotherapy In Standard Risk Medulloblastoma
Brief Title: Radiation Therapy Plus Combination Chemotherapy in Treating Children With Medulloblastoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000269521; SIOP-PNET-4; EU-20244; UKCCSG-CNS-2003-05
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2007-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood medulloblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Cisplatin; Lomustine; Vincristine; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: lomustine
Drug: vincristine sulfate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving radiation therapy in different ways with combination chemotherapy may kill any remaining tumor cells following surgery. It is not yet known which radiation therapy regimen combined with combination chemotherapy is more effective in treating medulloblastoma.

PURPOSE: Randomized phase III trial to compare different radiation therapy regimens plus combination chemotherapy in treating children who have undergone surgery for medulloblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the event-free survival rate in pediatric patients with standard-risk medulloblastoma treated with conventional vs hyperfractionated radiotherapy and vincristine followed by maintenance with cisplatin, lomustine, and vincristine.
* Compare the overall survival of patients treated with these regimens.
* Compare the pattern of relapse, especially local relapse (tumor bed or posterior fossa outside tumor bed), in patients treated with these regimens.
* Determine the toxicity of surgery and whether there are identifiable factors that correlate with toxicity in these patients.
* Determine the impact of any surgical complications on commencement of adjuvant therapy and event-free survival of these patients.
* Compare late sequelae, in terms of health status, endocrine deficiencies, and hearing loss, in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to country. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Within 28-40 days after surgical resection, patients undergo conventional fractionated radiotherapy once daily, 5 days a week, for 6-7 weeks. Patients also receive vincristine IV once weekly for 8 weeks.
* Arm II: Beginning as in arm I, patients undergo hyperfractionated radiotherapy twice daily, 5 days a week, for 6-7 weeks. Patients also receive vincristine as in arm I.
* Maintenance chemotherapy:Six weeks after completion of radiotherapy, all patients receive cisplatin IV over 6 hours and oral lomustine on day 1 and vincristine IV on days 1, 8, and 15. Treatment repeats every 6 weeks for 8 courses.

Patients are followed at least every 6 months for 3 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 316 patients (158 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed medulloblastoma, including the following variants:

  * Classic
  * Nodular/desmoplastic
  * Large cell
  * Melanotic
  * Medullomyoblastoma
* Prior total or subtotal surgical removal of tumor within the past 28-40 days

  * No more than 1.5 cm^2 residual tumor by early postoperative MRI or CT scan
* No brainstem or supratentorial primitive neuroectodermal tumor
* No atypical teratoid rhabdoid tumor
* No known predisposition to medulloblastoma (e.g., Gorlin's syndrome)
* No CNS metastasis (supratentorial, arachnoid of the posterior fossa, or craniospinal axis) by MRI
* No clinical evidence of metastasis outside the CNS
* No tumor cells in lumbar cerebrospinal fluid by cytospin

PATIENT CHARACTERISTICS:

Age

* 3 to 21

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Hematological function less than CTC grade 2

Hepatic

* Liver function less than CTC grade 2

Renal

* Renal function less than CTC grade 2

Other

* Not pregnant
* Fertile patients must use effective contraception
* Able to receive radiotherapy twice daily
* Vital functions within age-appropriate normal range
* Audiological function less than CTC grade 2
* No medical contraindication to radiotherapy or chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Concurrent dexamethasone as an antiemetic allowed, provided all other therapies have failed

Radiotherapy

* No concurrent cobalt irradiation

Surgery

* See Disease Characteristics

Other

* No prior treatment for brain tumor or any other malignancy

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 316 (Estimated)
Dates: Start 2003-02

PRIMARY OUTCOMES:
Comparison of event-free survival at 3 years

SECONDARY OUTCOMES:
Comparison of overall survival
Comparison of the pattern of relapse (i.e., local relapse [tumor bed and posterior fossa outside tumor bed])
Comparison of late sequelae, in terms of health status, quality of life, hearing loss, and endocrine deficiencies
Toxicity of neurosurgery

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta Lannering, MD, PhD, Study Chair — Ostra Sjukhuset
Locations (8):
- U.Z. Gasthuisberg, Leuven, Belgium
- Institut Curie Hopital, Paris, France
- Universitaets - Kinderklinik Wuerzburg, Würzburg, Germany
- Ospedale Infantile Regina Margherita, Turin, Italy
- Academisch Medisch Centrum at University of Amsterdam, Amsterdam, Netherlands
- Hospital de Cruces, Vizcaya, Spain
- Ostra Sjukhuset, Gothenburg, Sweden
- Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England, United Kingdom